CLINICAL TRIAL: NCT00977210
Title: A Phase I Trial of OXi4503 (a Vascular Disrupting Agent) Given by 3 Weekly Intravenous Infusions to Patients With Advanced Solid Tumors.
Brief Title: Safety Study of OXi4503 (a Vascular Disrupting Agent) Given by 3 x Weekly Intravenous Infusions to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH1/098
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Solid Tumors
Keywords: Phase 1; oxi4503; oxigene; cruk; solid tumors; VDA; vascular disrupting agent
MeSH Terms: interventions — Oxi 4503

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OXi4503 (Experimental)
  Interventions: Drug: OXi4503

INTERVENTIONS:
Drug: OXi4503 — OXi4503 will be administered weekly for 3 weeks followed by a week with no treatment. The starting dose will be 0.06 mg/m2 given as an intravenous infusion over 10 minutes.

SUMMARY:
The purpose of this study is to establish the Maximum Tolerated Dose (MTD) of OXi4503 given by weekly infusions to patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer.
* Written informed consent.
* Age >/= 18 years.
* Life expectancy of at least 12 weeks.
* World Health Organization (WHO) performance status of 0 or 1.
* Adequate Hematological and biochemical indices to support investigational therapy.
* All women of childbearing potential (WOCBP) must have a negative serum pregnancy test.
* WOCBP and fertile men and their partners must agree to use an effective form of contraception during the study and for 90 days after the last dose of study medication.
* Measurable and evaluable disease.
* All toxic manifestations of previous treatment must have resolved.
* Able to undergo MRI scanning.

Exclusion Criteria:

* Radiotherapy, endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosureas and Mitomycin-C) prior to treatment.
* Pregnant and lactating women.
* Major thoracic and/or abdominal surgery in the preceding four weeks from which the patient has not yet recovered.
* Patients which have active uncontrolled infections.
* Patients with any other condition that in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Patients known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Previous or ongoing cardiac conditions.
* Uncontrolled hypertension.
* Patients taking any drug known to prolong the QTc interval.
* Patients who have had any ischaemic or vascular damage from previous radiotherapy.
* Patients taking warfarin or heparin.
* Patients taking naproxen.
* Patients taking supplements or multivitamins containing vitamin C.
* Patients should not be taking any other investigational drug for the duration of the study.
* Patients with brain metastases or neurological tissue involvement of the spinal column.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To establish the Maximum Tolerated Dose (MTD) of OXi4503 given by weekly intravenous infusions. | 4 weeks

SECONDARY OUTCOMES:
To investigate the pharmacokinetic (PK) and pharmacodynamic (PD) behavior of OXi4503. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - CRUK Investigational Site, Manchester
  - CRUK Investigational Site, Middlesex

REFERENCES:
- [Derived] Patterson DM, Zweifel M, Middleton MR, Price PM, Folkes LK, Stratford MR, Ross P, Halford S, Peters J, Balkissoon J, Chaplin DJ, Padhani AR, Rustin GJ. Phase I clinical and pharmacokinetic evaluation of the vascular-disrupting agent OXi4503 in patients with advanced solid tumors. Clin Cancer Res. 2012 Mar 1;18(5):1415-25. doi: 10.1158/1078-0432.CCR-11-2414. Epub 2012 Jan 10. PMID 22235096